CLINICAL TRIAL: NCT03549403
Title: Effects of Patient-centered Pre- and Postoperative Telephone Education on the Experienced Health and Health-care Costs in Day Surgery by Adult Patients: A Randomized Controlled Trial.
Brief Title: Effects of Patient-centered Telephone Education in Day Surgery
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oulu (Other)
Collaborators: Oulu University Hospital (Other)
Responsible Party: Principal Investigator, Mira Rajala, McS, PhD-student, University Teacher, University of Oulu
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 152/2017
Record Dates: First submitted 2018-04-23; First posted 2018-06-08 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Health, Subjective; Cost Effectiveness
Keywords: Telephone education; Effectiveness; Health; Cost; Day surgery; Adult patient

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient-centered telephone education (Experimental): Patients receive the preoperative call home one week before the day surgery and postoperatively 3-8 days after the day surgery. On the day of surgery patients receive current education.
  Interventions: Behavioral: Patient-centered telephone education
- Current education practice (No Intervention): Patient´s education is implemented in accordance with current practice, where day surgery adult patients receive preoperative education over the phone one week prior to day surgery and postoperative education during on the day of surgery.

INTERVENTIONS:
Behavioral: Patient-centered telephone education — The intervention will be carried out in accordance with the guidelines and the contents of the patient-centered telephone education intervention in the same way with every patient. The education call duration is approximately 15 to 30 minutes.
  Arms: Patient-centered telephone education

SUMMARY:
This study describe and evaluate the effectiveness of patient-centered telephone education in day surgery. The aim is to evaluate the effects of patient-centered telephone education on the experienced health of adult patients and the costs of healthcare in day surgery. Telephone education intervention is planned in co-operation with the day surgery unit´s healthcare staff.

Half of participants will receive current education in day surgery, while the other half will receive developed patient-centered telephone education before and after day surgery.

DETAILED DESCRIPTION:
Research is an experimental randomized controlled trial -study and it will be carried out in a Finnish day surgery unit.

Research questions are as follows:

1. What are the implications of patient-centered pre- and postoperative telephone education for the experienced health of day surgery adult patients? Hypothesis 1: The experimental health of the trial group is better than the control group.
2. What is the impact of patient-centered pre- and postoperative telephone education on the costs of healthcare in day surgery adult patients? Hypothesis 1: The costs of healthcare in the trial group is lower than in the control group.

The aim is to produce new information that is used in the design and implementation of patient-centered and cost-effective patient education as well as develop patient education more patient-centered.

Patients are randomized to the trial (n = 60) and the control group (n = 60) in the order in which they receive the surgery time. The sample size is verified by force analysis.

Intervention group´s education: The nurse will call the preoperative call to the patient home one week before the day surgery and postoperatively within 3-8 days after the day surgery. The intervention will be carried out in accordance with the guidelines and the contents of the developed patient-centered telephone education intervention in the same way in each patient. The call duration is approximately 15 to 30 minutes. Telephone education is carried out by a nurse responsible for preoperative telephone education in day surgery unit and 2-3 anesthesia nurses who have also participated in the intervention planning. The researcher provides them with guidance on patient-centered telephone education prior to intervention.

Control group´s education: The control group's education is carried out by nurses responsible for patient education in the day surgery unit who have not been involved in the planning and implementation of the intervention. Education is implemented in accordance with current practice, where day surgery adult patients receive preoperative education over the phone one week prior to day surgery and postoperative education during the day surgery.

The collection of the data is done by the modified Oldwellactive Oulu -instrument, whose reliability has been found to be acceptable in the previous studies.The preliminary questionnaire is sent before surgery to the patient and returns the questionnaire is upon arrival in the day surgery. Nurses receive the questionnaires and put them in a sealed mailbox placed in the department. The investigator is responsible for clearing the mailbox. The questionnaire for the final measurement is given by nurses to the day surgery patient in connection with discharge education. The questionnaire is requested to fill in two weeks after the surgery and return it with a supplied postage stamped addressed envelope.

The costs of health-care are calculated in the number and duration of postoperative patient´s phone calls to the day surgery unit of the patient documents as well as separate book counts. Additionally calculated the number of emergency / polyclinic / hospital department visits and laboratory examinations / X-ray images after the day surgery of patient documents for 3 months. The costs of the trial group are compared to the control group before and after the surgery.

Patient randomization is performed by various nurses than by the intervention itself, thus avoiding the risk of selective randomization. A randomizing nurse will share day surgery adult patients meeting the criteria for entry into the trial and control groups in the order in which they receive the surgery time. Patients are provided with a Register Statement and an identification code list to ensure the intervention´s planned implementation of the study. The Register Statement of the patients is stored on the researcher's computer behind the password. Questionnaires are encoded that the identity of the patients is not disclosed. In the health-care cost´s calculation, markings from patient documents are processed without personal identifiers, so the issues being processed can not be combined with a particular patient.

Questionnaires are stored in a locked locker and all material on the researcher's computer behind the password. The researcher is responsible for the retention and proper disposal of the material, questionnaires, registration descriptions and identification code lists. Research findings are set to scientific criticism at the publishing stage and possible criticism is taken into account. The results are not generalized or prettify. Reporting aims at open, clear and accurate.

The data is analyzed using descriptive parameters and regression analysis for preliminary and final status by testing the difference between the trial and control groups by the Mann-Whitney U-test. The Consort checklist is used to evaluate and report the intervention implementation.

ELIGIBILITY:
Inclusion Criteria:

* arrive at the surgery from home
* leave latest at the next morning of the surgery
* leave home after surgery
* is 18-64 years old
* be able to respond to the questionnaire independently.

Exclusion Criteria:

* over 65 years old patients
* patients who need institutional care after surgery
* patients who arrive to surgery from a institutional care unit

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Experienced health | Up to two weeks after surgery
  The questionnaire assess the impact of patient-centered telephone education to the day surgery patients´ experienced health, such as mobility, sleep, normal functions of survival, intellectual activities, ailments and symptoms, anxiety and energetic aspects.
Health-care costs | Up to three months after surgery
  Patient-centered telephone education´s measures to the number of patient´s postoperative treatment

CONTACTS AND LOCATIONS:
Overall Officials: Maria Kääriäinen, PhD, Study Director — University of Oulu
Locations (1):
- University of Oulu, Oulu, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rajala M, Kaakinen P, Fordell M, Kaariainen M. The Quality of Patient Education in Day Surgery by Adult Patients. J Perianesth Nurs. 2018 Apr;33(2):177-187. doi: 10.1016/j.jopan.2016.02.013. Epub 2017 Mar 30. PMID 29580597